CLINICAL TRIAL: NCT06724029
Title: Neurosurgical Outcome Network Per La Predizione Dell'outcome in Neurochirurgia
Brief Title: Neurosurgical Outcome Network
Acronym: NEON
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: NEON
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Aneurysms; Arteriovenous Malformations; Cavernomas; Skull Base Tumors; Moyamoya Disease; Dural Fistulas; Subdural Hematoma; Extradural Hematoma; Subarachnoid Hemorrhage; Hydrocephalus; Parkinson's Disease; Spasticity; Trigeminal Neuralgia; Craniofacial Pain; Neuropathic Pain; Tremor; Dystonias; Obsessive-compulsive Disorder; Drug-resistant Epilepsy; Depression; Normal Pressure Hydrocephalus; Tumors of Peripheral Nerves; Chiari Malformation Type 1
Keywords: Neurosurgery Outcome Artificial Intelligence predictors
MeSH Terms: conditions — Aneurysm; Arteriovenous Malformations; Moyamoya Disease; Hematoma, Subdural; Hematoma, Epidural, Spinal; Subarachnoid Hemorrhage; Hydrocephalus; Muscle Spasticity; Trigeminal Neuralgia; Facial Pain; Neuralgia; Tremor; Dystonic Disorders; Obsessive-Compulsive Disorder; Drug Resistant Epilepsy; Depression; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The evaluation of neurosurgical outcomes varies from center to center, and the predictive factors that determine these outcomes are not fully known or shared. This study aims to assess outcomes and their predictors using measures agreed upon by the participating centers. Standardizing the evaluation of outcomes and predictors improves the quality of research, allows for data comparison, and facilitates a "common language" in routine clinical practice. Most importantly, it influences therapeutic decisions in various neurosurgical conditions. Clinically, the identified predictors can also be used during preoperative assessments to provide more precise guidance to patients undergoing surgery.

DETAILED DESCRIPTION:
The evaluation of outcome indicators, quality of life, and complexity in Neurosurgery has gained significant importance not only at a clinical and therapeutic level but also as a tool to assess the effectiveness and efficiency of the healthcare system. This study aims to evaluate neurosurgical outcomes and their predictors using measures shared among participating centers. Such evaluation varies from center to center, and the predictive factors are not entirely known or shared. Standardizing the evaluation of outcomes and predictors improves research quality, enables data comparison, and fosters a common language in everyday clinical practice. Most importantly, it influences therapeutic decisions in various neurosurgical pathologies.

Primary Objective: Collect and describe the pre- and postoperative clinical, cognitive, and psychological status in various neurosurgical pathologies.

Secondary Objectives: Identify outcome predictors. Primary Endpoint: Description of pre- and postoperative clinical, cognitive, and psychological data of patients undergoing neurosurgical intervention.

Secondary Endpoints: Analyze the association between preoperative indicators collected and postoperative outcomes. Specific predictors and outcome measures for each neurosurgical pathology will be considered and reported in Appendix 1. Patient enrollment from Neurosurgery Departments; collection of clinical, cognitive, and psychological data before the intervention and during follow-up after the intervention (timing varies depending on the neurosurgical pathology); data analysis through AI. For all neurosurgical pathologies, the following data will be collected: sociodemographic, clinical (Charlson Comorbidity Index, heart disease, diabetes, Chronic Obstructive Pulmonary Disease, hypertension, Body Mass Index, smoking, psychiatric pathology, admission date, intervention date, discharge date, Modified Rankin Scale, American Society of Anesthesiologists, weight, height), anesthesiological (collected only by FINCB), and complication-related data (Novel Therapy-Disability-Neurology).

ELIGIBILITY:
Inclusion Criteria:

* Neuro-oncological pathology: supratentorial and subtentorial tumors, intra and extra axial tumors excluding the skull base (anterior, middle and posterior fossa; sellar and parasellar region)
* Basicranial pathology: tumors originating from the anterior cranial fossa, middle cranial fossa and posterior cranial fossa, sellar region with or without supratentorial/parasellar development.
* Vascular pathology: aneurysms, AVMs, cavernomas, other pathologies (Moyamoya disease, dural fistulas, nontraumatic hematomas)
* Traumatic pathology: diffuse damage (nonvisible diffuse damage, diffuse damage, diffuse damage with edema, diffuse damage with shift) and focal damage (acute/subacute/chronic subdural hematoma, extradural hematoma, subarachnoid hemorrhage, intraparenchymal hematoma, fractures); hydrocephalus. The inclusion criterion for chronic subdural hematoma is recent bleeding for TBI with CT finding of chronic subdural hematoma candidate for evacuation surgery.
* Spinal pathology: degenerative cervical (anterior/posterior), myelopathic, and trauma pathology; instrumented, uninstrumented thoracolumbar pathology (disc pathology, canal pathology), and trauma pathology; oncologic spinal pathology.
* Functional pathology: Parkinson's disease, spasticity, trigeminal neuralgia, craniofacial pain/algia, neuropathic pain, tremor, dystonias, obsessive compulsive disorder, drug-resistant epilepsies, depression. Normotensive hydrocephalus.
* Peripheral nervous system pathology: peripheral nerve compression syndromes, peripheral nerve and plexus tumors, brachial plexus and peripheral nerve trauma (contusion and section)
* Malformative pathology: Chiari malformation type 1 and craniostenoses including both those framed in malformative syndromes and those not framed in malformative syndromes (monosutural craniostenoses: trigonocephaly, plagiocephaly, scaphocephaly; multisutural craniostenoses). Malformative hydrocephalus.
* For cognitive and psychological assessment: age 18 years or older; adequate understanding of Italian language; diagnosis of glioma, meningioma, vascular pathology, spinal pathology

Exclusion Criteria:

* For cognitive and psychological assessment: patients with psychiatric diseases in history and/or taking psychotropic drugs; presence of overt cognitive decline (not due to the injury) in history; patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, with neurosurgical pathology
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Collect data | 5 years
  Collect and describe the pre- and postoperative clinical status in various neurosurgical pathologies.
Collection data | 5 years
  Collect and describe the pre- and postoperative cognitive status in various neurosurgical pathologies.
Collection data | 5 years
  Collect and describe the pre- and postoperative psychological status in various neurosurgical pathologies.

SECONDARY OUTCOMES:
Identify Predictors | 1 year
  Identify outcome predictors.

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - 1. ASST Papa Giovanni XXIII, Bergamo, BG
  - Spedali Civili Brescia, Brescia, BS
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia, BS
  - Ospedale Moriggia Pelascini, Gravedona, Como
  - ASST Lariana, Ospedale S. Anna, Como, CO
  - ASST Cremona, Cremona, CR
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - ASST della Valtellina ed Alto Lario, Sondrio, SO
  - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale F. Spaziani di Frosinone, Frosinone
  - Ospedale Alessandro Manzoni, Lecco
  - ASST Ovest Milanese, Legnano
  - Ospedali Riuniti di Livorno -Azienda USL Toscana nord ovest, Livorno
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Santi Paolo e Carlo, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Istituto Clinico Città Studi, Milan
  - Policlinico di Monza, Monza
  - A.R.N.A.S. Ospedali Civico di Palermo, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - ASL Roma 1, Roma
  - Fondazione Policlinico Universitario Gemelli di Roma, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Azienda Sanitaria Universitaria Friuli Centrale di Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terrapon APR, Zattra CM, Voglis S, Velz J, Vasella F, Akeret K, Held U, Schiavolin S, Bozinov O, Ferroli P, Broggi M, Sarnthein J, Regli L, Neidert MC. Adverse Events in Neurosurgery: The Novel Therapy-Disability-Neurology Grade. Neurosurgery. 2021 Jul 15;89(2):236-245. doi: 10.1093/neuros/nyab121. PMID 33887774
- [Background] RANKIN J. Cerebral vascular accidents in patients over the age of 60. II. Prognosis. Scott Med J. 1957 May;2(5):200-15. doi: 10.1177/003693305700200504. No abstract available. PMID 13432835
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Grinnon ST, Miller K, Marler JR, Lu Y, Stout A, Odenkirchen J, Kunitz S. National Institute of Neurological Disorders and Stroke Common Data Element Project - approach and methods. Clin Trials. 2012 Jun;9(3):322-9. doi: 10.1177/1740774512438980. Epub 2012 Feb 27. PMID 22371630
- [Background] Jakola AS, Unsgard G, Solheim O. Quality of life in patients with intracranial gliomas: the impact of modern image-guided surgery. J Neurosurg. 2011 Jun;114(6):1622-30. doi: 10.3171/2011.1.JNS101657. Epub 2011 Feb 11. PMID 21314270
- [Background] Sagberg LM, Drewes C, Jakola AS, Solheim O. Accuracy of operating neurosurgeons' prediction of functional levels after intracranial tumor surgery. J Neurosurg. 2017 Apr;126(4):1173-1180. doi: 10.3171/2016.3.JNS152927. Epub 2016 Jun 17. PMID 27315026
- [Background] Weldring T, Smith SM. Patient-Reported Outcomes (PROs) and Patient-Reported Outcome Measures (PROMs). Health Serv Insights. 2013 Aug 4;6:61-8. doi: 10.4137/HSI.S11093. eCollection 2013. PMID 25114561
- [Background] Tomlinson SB, Piper K, Kimmell KT, Vates GE. Preoperative Frailty Score for 30-Day Morbidity and Mortality After Cranial Neurosurgery. World Neurosurg. 2017 Nov;107:959-965. doi: 10.1016/j.wneu.2017.07.081. Epub 2017 Jul 20. PMID 28736345
- [Background] Reponen E, Tuominen H, Korja M. Evidence for the use of preoperative risk assessment scores in elective cranial neurosurgery: a systematic review of the literature. Anesth Analg. 2014 Aug;119(2):420-432. doi: 10.1213/ANE.0000000000000234. PMID 25046789